CLINICAL TRIAL: NCT02716584
Title: Physical Exercise Effects on Determinants of Social Integration in Schizophrenia
Brief Title: Benefits of Physical Exercise in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2026-P; 1I21RX002026 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-03-23 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Exercise; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical exercise (Experimental): Participants participate in brisk walking exercises.
  Interventions: Behavioral: Physical exercise
- Stretching exercise (Active Comparator): Participants participate in non-aerobic, non-Yoga stretching exercises
  Interventions: Behavioral: Stretching exercise

INTERVENTIONS:
Behavioral: Physical exercise — Veterans in the physical exercise group will participate in a 12-week, instructor-led, outdoor brisk walking exercise program conducted in small groups, held 3 times per week, gradually increasing walking time until reaching a maximum of 40-minutes per session. The heart rate of each Veteran will be monitored during the walking sessions to help ensure maintenance of a target peak heart rate of 60% to 70% of the maximum for the individual's age (i.e., 220-age).
  Arms: Physical exercise
Behavioral: Stretching exercise — Veterans in the control condition will participate in instructor-led, non-aerobic stretching exercises conducted in small groups, held 3 times per week.
  Arms: Stretching exercise

SUMMARY:
Impairments in social integration, characterized by low marriage rates, few friendships, and a high frequency of living alone, affect the vast majority of Veterans with schizophrenia. The primary aim of this proposal is to test the efficacy of a novel rehabilitation treatment approach, engaging in physical exercise, at improving two determinants of social integration which are impaired in schizophrenia: cognition and affect.

DETAILED DESCRIPTION:
Difficulties in social integration pose a major mental health problem for Veterans with schizophrenia. Reviews of the literature indicate that Veterans with schizophrenia have lower marriage rates, fewer friendships, and higher rates of living alone than the general population. Poor social integration is also associated with early mortality. To gain traction on this problem, it will be necessary to find treatments that address key determinants of social integration. Evidence indicates that impairments in cognition and affect are among the key determinants of this area of functioning. Findings from the broader rehabilitation literature support a novel conceptual approach to this problem, namely engagement in physical exercise. Physical exercise is associated with improvements in attention, episodic memory, working memory, speed of processing, and executive control. In addition, physical exercise is associated with increases in positive affect and decreases in negative affect. Findings on the effects of physical exercise on cognition and affect have been reported for normal aging, mild cognitive impairment, neurodegenerative disorders, oncology, and depression, but is an area of investigation relatively new to schizophrenia. The proposed study will include 54 Veterans with schizophrenia or schizoaffective disorder (aged 45-65) who will be matched on baseline levels of cardiorespiratory fitness, and then randomized (2:1) to a walking exercise group (n=36) or a control comparison group (n=18). Veterans in the exercise group will participate in a 12-week, instructor-led, outdoor brisk walking exercise program conducted in small groups (n=6), held 3 times per week, gradually increasing walking time until reaching a maximum of 40-minutes per session. The heart rate of each Veteran will be monitored during the walking sessions to help ensure maintenance of a target peak heart rate of 60% to 70% of the maximum for the individual's age (i.e., 220-age). Veterans in the control group will participate in instructor-led, non-aerobic stretching exercises in small groups (n=6) with the duration, frequency, and total number of sessions matched to the exercise group. Primary outcome measures of cardiorespiratory fitness, cognition, and positive and negative affect of participants in both groups will be measured at baseline and the 12-week end-point assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual (DSM) - 5 diagnosis of schizophrenia or schizoaffective disorder;
* age 40-65;
* screened for physical health risks (i.e., no serious heart condition, dizziness, bone or joint problems posing safety concerns, ambulatory limitations);
* clinically stable (e.g., no inpatient hospitalizations for 3 months prior to enrollment; no change in type of antipsychotic medication in the past 4 weeks)

Exclusion Criteria:

* evidence of alcohol or substance use disorder (moderate or greater severity) per DSM-5 criteria in the past 3 months;
* clinically significant neurological disease as determined by medical history (e.g., seizure disorder);
* history of serious head injury with loss of consciousness >1 hour;
* participation in an exercise program within past 6 months;
* not able to understand spoken and written English sufficiently to comprehend consent procedures.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Kern, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and SAP will be available one year after study completion and will be available indefinitely.
Access Criteria: The study protocol and SAP will be available to the public domain.

REFERENCES:
- [Background] Malchow B, Reich-Erkelenz D, Oertel-Knochel V, Keller K, Hasan A, Schmitt A, Scheewe TW, Cahn W, Kahn RS, Falkai P. The effects of physical exercise in schizophrenia and affective disorders. Eur Arch Psychiatry Clin Neurosci. 2013 Sep;263(6):451-67. doi: 10.1007/s00406-013-0423-2. Epub 2013 Jul 20. PMID 23873090
- [Background] Knochel C, Oertel-Knochel V, O'Dwyer L, Prvulovic D, Alves G, Kollmann B, Hampel H. Cognitive and behavioural effects of physical exercise in psychiatric patients. Prog Neurobiol. 2012 Jan;96(1):46-68. doi: 10.1016/j.pneurobio.2011.11.007. Epub 2011 Nov 24. PMID 22120173
- [Background] Kimhy D, Vakhrusheva J, Bartels MN, Armstrong HF, Ballon JS, Khan S, Chang RW, Hansen MC, Ayanruoh L, Lister A, Castren E, Smith EE, Sloan RP. The Impact of Aerobic Exercise on Brain-Derived Neurotrophic Factor and Neurocognition in Individuals With Schizophrenia: A Single-Blind, Randomized Clinical Trial. Schizophr Bull. 2015 Jul;41(4):859-68. doi: 10.1093/schbul/sbv022. Epub 2015 Mar 23. PMID 25805886
- [Background] Heggelund J, Kleppe KD, Morken G, Vedul-Kjelsas E. High aerobic intensity training and psychological States in patients with depression or schizophrenia. Front Psychiatry. 2014 Oct 30;5:148. doi: 10.3389/fpsyt.2014.00148. eCollection 2014. PMID 25400592
- [Background] Pajonk FG, Wobrock T, Gruber O, Scherk H, Berner D, Kaizl I, Kierer A, Muller S, Oest M, Meyer T, Backens M, Schneider-Axmann T, Thornton AE, Honer WG, Falkai P. Hippocampal plasticity in response to exercise in schizophrenia. Arch Gen Psychiatry. 2010 Feb;67(2):133-43. doi: 10.1001/archgenpsychiatry.2009.193. PMID 20124113

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Exercise | Stretching Exercise
Started | 35 | 18
Completed | 27 | 13
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Exercise | Stretching Exercise | Total
Number analyzed (Participants) | 35 | 18 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (6.2) | 55.7 (7.1) | 56.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 33 | 18 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 12 | 35
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Participants were all Veterans.
  participants
    United States | 35 | 18 | 53
VO2max [Mean (Standard Deviation); unit: ml.kg-1.min-1] | 22.6 (15.3) | 23.3 (12.4) | 22.8 (14.3)
Birchwood Social Functioning Scale [Mean (Standard Deviation); unit: units on a scale] — Birchwood Social Functioning Scale - This scale is a measure of social functioning that includes seven domains (social engagement, interpersonal communication, independence - performance, independence - competence, recreation, prosocial behavior, and employment). The subscale scores are summed to yield a total score. The primary outcome measure is a total score with a possible range from 0 to 223; higher scores represent better social functioning.
  units on a scale | 121.0 (24.7) | 116.7 (22.1) | 119.5 (23.7)

OUTCOME MEASURES:

1. Primary Outcome: VO2max
Description: Measure of aerobic capacity (VO2max) is derived by using a regression formula based on age, weight, sex, and time to complete walking of one mile. Because scores are derived using a regression equation, there is no absolute minimum or maximum value; higher scores represent better aerobic capacity.
Time Frame: Change from baseline to 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: ml.kg-1.min-1
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
ml.kg-1.min-1 | 4.0 (4.0) | 0.2 (5.6)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Data were analyzed using a 2 (groups) x 2 (time: baseline, endpoint) repeated measures ANCOVA with number of exercise sessions attended as a covariate; Test type: Superiority; p = 0.02, ANCOVA; Effect size = 0.41

2. Primary Outcome: Total Score for Social Functioning
Description: Birchwood Social Functioning Scale is a measure of social functioning. The total score for social functioning is calculated by summing the raw scores from each of the seven subscales (social engagement, interpersonal communication, independence - performance, independence - competence, recreation, prosocial behavior, employment); possible range is 0 to 223 with higher scores representing better social functioning.
Time Frame: Change from baseline to 12 week endpoint assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
score on a scale | 3.7 (10.9) | -2.5 (10.2)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.06, ANCOVA; Data were analyzed using a 2 (groups) x 2 (time: baseline, endpoint) repeated measures ANCOVA with number of sessions attended as a covariate; Effect size = 0.35

3. Primary Outcome: Total Score for Speed of Processing (i.e., Cognition) as Assessed by the Brief Assessment of Cognition in Schizophrenia (BACS) Symbol Coding Test
Description: Brief Assessment of Cognition in Schizophrenia (BACS) is a measure of speed of information processing. The total score for speed of processing (i.e., cognition) is calculated by summing the number of symbol-code pairs completed correctly on the BACS Symbol Coding test within the allotted 90 second time limit. Scores range from 0 to 110 with higher scores representing better information processing speed.
Time Frame: Change from baseline to 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
score on a scale | -0.4 (4.9) | 2.3 (5.4)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.13, ANCOVA; [statistical method as in outcome 2, analysis 1]

4. Primary Outcome: Total Score for Positive Affect as Assessed by the Positive and Negative Affect Scale (PANAS)
Description: Positive and Negative Affect Scale is a measure of an individual's positive and negative affect. The scale includes 32 items; 16 denote positive affect and 16 denote negative affect. Each item is rated on a scale of 1 (very slightly or not at all) to 5 (extremely). The total score for PANAS positive affect is calculated by summing the ratings for items denoting positive affect. Scores range from 16 to 80; higher scores represent better positive affect.
Time Frame: Change from baseline to the 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
score on a scale | -5.6 (12.6) | -8.9 (14.1)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.73, ANCOVA — The analyses for cohorts 1 and 2 utilized the a priori endpoint assessment conducted 1-2 weeks after completion of training; The data were analyzed using a 2 (groups) x 2 (time: baseline, endpoint) repeated measures ANCOVA with number of sessions attended as a covariate; Effect size = .19
Statistical Analysis 2: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = .33, ANCOVA — For cohort 3, positive affect was measured at baseline and a midpoint assessment; The data were analyzed using a 2 (groups) x 2 (time: baseline, midpoint) repeated measures ANCOVA with number of sessions attended as a covariate; Effect size = 0.73

5. Primary Outcome: Total Score for Negative Affect as Assessed by the Positive and Negative Affect Scale (PANAS)
Description: Positive and Negative Affect Scale is a measure of an individual's positive and negative affect. The scale includes 32 items; 16 denote positive affect and 16 denote negative affect. Each item is rated on a scale of 1 (very slightly or not at all) to 5 (extremely). The total score for PANAS negative affect is calculated by summing the ratings for items denoting negative affect. Scores range from 16 to 80; lower scores represent better levels of negative affect.
Time Frame: Change from baseline to the 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
score on a scale | 3.8 (8.8) | 2.6 (6.5)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.62, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Effect size = -0.21
Statistical Analysis 2: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = .23, ANCOVA — For cohort 3, positive affect was measured at a baseline and midpoint assessment; [statistical method as in outcome 4, analysis 2]; Effect size = 0.77

6. Primary Outcome: Composite Score From Non-social Cognition Battery
Description: Raw scores (i.e., total scores) for the following tests will be transformed to z-scores: attention (CPT-IP), speed of processing (BACS symbol coding), working memory (WAIS-IV letter-number sequencing test), verbal learning (Hopkins Verbal Learning Test - Revised), and executive control (AX-CPT). The outcome measure is the mean z-score. The composite z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean of the overall sample of study participants. Negative numbers indicate values lower than other study participants and positive numbers indicate values higher than other study participants.
Time Frame: Change from baseline to the 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
z-score | .01 (.50) | .06 (.52)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.57, ANCOVA; [statistical method as in outcome 2, analysis 1]; Effect size = 0.02

7. Secondary Outcome: Composite Score From Social Cognition Battery
Description: Raw scores (i.e., total scores) for the following tests will be transformed to z-scores: emotion perception (Facial Emotion Identification Test), social perception (Half-Profile of Nonverbal Sensitivity; PONS), theory of mind (The Awareness of Social Inference Test; TASIT - Part 2), empathy (empathic accuracy test). The outcome measure is the mean z-score. The composite z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean of the overall sample of study participants. Negative numbers indicate values lower than other study participants and positive numbers indicate values higher than other study participants.
Time Frame: Change from baseline to the 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
z-score | .06 (.46) | -.17 (.47)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.12, ANCOVA; [statistical method as in outcome 2, analysis 1]; Effect size = 0.35

8. Secondary Outcome: BDNF Value
Description: BDNF concentration will be quantified by enzyme-linked immunosorbent assay (R&D Systems). The value will be expressed in ng/ml.
Time Frame: Change from baseline to the 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
ng/ml | -1.04 (9.57) | -7.31 (8.01)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.07, ANCOVA; [statistical method as in outcome 2, analysis 1]; Effect size = 0.72

9. Secondary Outcome: Positive Symptom Subscale Score From the BPRS
Description: The Brief Psychiatric Rating Scale (BPRS) is a measure of psychiatric symptom severity and includes subscale scores for positive and negative symptoms. The outcome score for positive symptoms is calculated by summing the ratings for items measuring hallucinations, unusual thought content, and conceptual disorganization; each item is rated on a scale of 1 to 7 with higher scores indicating greater symptom severity; possible range for positive symptoms is 0 to 21 with higher scores representing greater severity of positive symptoms.
Time Frame: Change from baseline to the 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
score on a scale | -1.2 (4.5) | -1.2 (1.5)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.88, ANCOVA; [statistical method as in outcome 2, analysis 1]; Effect size = 0.00

10. Secondary Outcome: Negative Symptom Subscale Score From the BPRS
Description: The Brief Psychiatric Rating Scale (BPRS) is a measure of psychiatric symptom severity and includes subscale scores for positive and negative symptoms. The outcome score for negative symptoms is calculated by summing the ratings for items measuring blunted affect, emotional withdrawal, and motor retardation; each item is rated on a scale of 1 to 7 with higher scores indicating greater symptom severity; possible range for negative symptoms is 0 to 21 with higher scores representing greater severity of negative symptoms.
Time Frame: Change from baseline to the 12-week endpoint assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Exercise | Stretching Exercise
Number analyzed (Participants) | 27 | 13
score on a scale | 0.1 (2.5) | 0.1 (2.8)
Statistical Analysis 1: Comparison: Physical Exercise vs Stretching Exercise; Test type: Superiority; p = 0.86, ANCOVA; [statistical method as in outcome 2, analysis 1]; Effect size = 0.05

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Physical Exercise | Stretching Exercise
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/18
Other Adverse Events (participants affected / at risk) | 0/35 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT02716584/Prot_SAP_000.pdf